CLINICAL TRIAL: NCT03854409
Title: An Open-label, Single- and Multiple-dose, Pharmacokinetic, Safety, and Tolerability Trial of Aripiprazole Long-acting Injectable Administered in the Deltoid or Gluteal Muscle in Adult Subjects With Schizophrenia or Bipolar I Disorder
Brief Title: A Trial of Single- and Multiple-doses of Aripiprazole in Adult Subjects With Schizophrenia or Bipolar I Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry); H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 031-201-00279
Record Dates: First submitted 2019-02-12; First posted 2019-02-26 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-12

CONDITIONS: Schizophrenia; Bipolar I Disorder
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A - Deltoid Site: Single Dose Group (Experimental): Participants will receive a single dose of aripiprazole LAI.
  Interventions: Drug: Aripiprazole
- Part A - Gluteal Site: Single Dose Group (Experimental): Participants will receive a single dose of aripiprazole LAI.
  Interventions: Drug: Aripiprazole
- Part A - Deltoid Site: Multiple Dose Group (Experimental): Participants will receive five injections of aripiprazole LAI, administered at monthly intervals.
  Interventions: Drug: Aripiprazole
- Part A - Gluteal Site: Multiple Dose Group (Experimental): Participants will receive five injections of aripiprazole LAI, administered at monthly intervals.
  Interventions: Drug: Aripiprazole
- Part B - Gluteal Site: Group 1 (X) (Experimental): Participants will receive a single dose of aripiprazole LAI.
  Interventions: Drug: Aripiprazole
- Part B - Gluteal Site: Group 1 (Y) (Experimental): Participants will receive a single dose of aripiprazole LAI.
  Interventions: Drug: Aripiprazole
- Part B - Gluteal Site: Group 2 (Experimental): Participants will receive a single dose of aripiprazole LAI.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Injection.
  Other Names: (OPC-14597)

SUMMARY:
The primary objective of this trial is to evaluate the pharmacokinetics (PK) of aripiprazole long-acting injectable (LAI) (420 mg) following deltoid or gluteal muscle administration in adult subjects with schizophrenia or bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 64 years of age, inclusive.
* Body mass index of 18 to 35 kg/m2, inclusive.
* A current diagnosis of schizophrenia or a current diagnosis of bipolar I disorder as defined by DSM-5 criteria.
* Prior history of tolerating aripiprazole per investigator's judgment.

Exclusion Criteria:

* Subjects who have met DSM-5 criteria for substance dependence within the past 180 days
* Use of any psychotropic medications other than their current non-aripiprazole antipsychotic or mood stabilizer(s) medication or subjects who use more than one antipsychotic or mood stabilizer(s) medication at screening.
* Subjects may not receive varenicline beyond screening.
* Use of any prescription medication not specifically approved by the medical monitor.
* Females who are pregnant or lactating. A negative serum pregnancy test must be confirmed prior to the first dose of IMP for all female subjects.
* Subjects who had participated in any clinical trial involving a psychotropic medication within 1 month prior to enrollment; subjects who had participated in a previous aripiprazole LAI trial within the last 1 year (ie, enrolled but did not receive aripiprazole LAI); or who had previously enrolled and received IMP in an aripiprazole LAI clinical trial.
* Any major surgery within 30 days prior to enrollment or scheduled/elective surgery during the trial.
* Subjects currently in an acute relapse of schizophrenia.
* Subjects with a current DSM-5 diagnosis other than schizophrenia or bipolar I disorder
* Electroconvulsive therapy must not be conducted within 2 months prior to administration of the IMP
* Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia as assessed by the investigator.
* History of or current hepatitis or acquired immunodeficiency syndrome or carriers of HBsAg, anti-HCV, and/or HIV antibodies.
* History of any significant drug allergy or known or suspected hypersensitivity, in particular to aripiprazole or other quinolinones.
* Subjects deemed intolerant of receiving injections.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Part A - Single Dose Group: Maximum Observed Plasma Concentration (Cmax) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 126
Part B - Group 1: Maximum Observed Plasma Concentration (Cmax) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part B - Group 2: Maximum Observed Plasma Concentration (Cmax) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part A - Single Dose Group: Plasma Concentration at 28 Days Postdose (C28) for Aripiprazole and Dehydro-Aripiprazole | Day 28
Part B - Group 1: Plasma Concentration at 28 Days Postdose (C28) for Aripiprazole and Dehydro-Aripiprazole | Day 28
Part B - Group 2: Plasma Concentration at 28 Days Postdose (C28) for Aripiprazole and Dehydro-Aripiprazole | Day 28
Part A - Single Dose Group: Time to Reach the Maximum Plasma Concentration (Tmax) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 126
Part B - Group 1: Time to Reach the Maximum Plasma Concentration (Tmax) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part B - Group 2: Time to Reach the Maximum Plasma Concentration (Tmax) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part A - Single Dose Group: Area Under the Concentration-Time Curve from time Zero to Time t (the Last Observable Concentration; AUCt) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 126
Part B - Group 1: Area Under the Concentration-Time Curve from time Zero to Time t (the Last Observable Concentration; AUCt) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part B - Group 2: Area Under the Concentration-Time Curve from time Zero to Time t (the Last Observable Concentration; AUCt) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part A - Single Dose Group: Area Under the Concentration-Time Curve from Time Zero to 28 Days Postdose (AUC0-28) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 28
Part B - Group 1: Area Under the Concentration-Time Curve from Time Zero to 28 Days Postdose (AUC0-28) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 28
Part B - Group 2: Area Under the Concentration-Time Curve from Time Zero to 28 Days Postdose (AUC0-28) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 28
Part A - Single Dose Group: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Aripiprazole (AUC∞) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 126
Part B - Group 1: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Aripiprazole (AUC∞) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part B - Group 2: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Aripiprazole (AUC∞) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part A - Single Dose Group: Terminal Phase Elimination Half-life (T1/2) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 126
Part B - Group 1: Terminal Phase Elimination Half-life (T1/2) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part B - Group 2: Terminal Phase Elimination Half-life (T1/2) for Aripiprazole and Dehydro-Aripiprazole | Day 1 to Day 57
Part A - Single Dose Group: Oral Clearance (CL/F) for Aripiprazole Only | Day 1 to Day 126
  Apparent clearance of the drug from plasma after extravascular administration (CL/F).
Part B - Group 1: Oral Clearance (CL/F) for Aripiprazole Only | Day 1 to Day 57
  Apparent clearance of the drug from plasma after extravascular administration (CL/F).
Part B - Group 2: Oral Clearance (CL/F) for Aripiprazole Only | Day 1 to Day 57
  Apparent clearance of the drug from plasma after extravascular administration (CL/F).
Part A - Multiple Dose Group: Maximum Observed Plasma Concentration (Cmax) for Aripiprazole and Dehydro-Aripiprazole (Following the Fifth Dose Only) | Day 113 to Day 169
  Fifth dose will be administered on Day 113.
Part A - Multiple Dose Group: Plasma Concentration at 28 Days Postdose (C28) for Aripiprazole and Dehydro-Aripiprazole | Day 29, Day 57, Day 84, Day 113, Day 141 (All post-dose)
Part A - Multiple Dose Group: Time to Reach the Maximum Plasma Concentration (Tmax) (Following the Fifth Dose Only) for Aripiprazole and Dehydro-Aripiprazole | Day 113 to Day 169
  Participants will receive their 5th dose on Day 113.
Part A - Multiple Dose Group: Area Under the Concentration-Time Curve from Time Zero to 28 Days Postdose (AUC0-28) (Following the Fifth Dose Only) for Aripiprazole and Dehydro-Aripiprazole | Day 113 to Day 169
  Participants will receive their 5th dose on Day 113.
Part A - Multiple Dose Group: Terminal Phase Elimination Half-life (T1/2) (Following the Fifth Dose Only) for Aripiprazole and Dehydro-Aripiprazole | Day 113 to Day 169
  Participants will receive their 5th dose on Day 113.
Part A - Multiple Dose Group: Oral Clearance (CL/F) (Following the Fifth Dose Only; for Aripiprazole Only) | Day 113 to Day 169
  Participants will receive their 5th dose on Day 113.
Part A - Multiple Dose Group: Ratio of Dehydro-Aripiprazole to Aripiprazole C28 and AUC0-28 (Following the Fifth Dose Only) | Day 113 (following fifth dose) to Day 141
  Participants will receive their 5th dose on Day 113.

SECONDARY OUTCOMES:
Part A - Single Dose: Number of Participants with an Adverse Event (AE) | Day 1 to End of Trial (Maximum 126 Days from First Dose)
  An AE is defined as any untoward medical occurrence in a clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Part A - Multiple Dose: Number of Participants with an Adverse Event (AE) | Day 1 to End of Trial (Maximum 169 Days from First Dose)
  An AE is defined as any untoward medical occurrence in a clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Part B: Number of Participants with an Adverse Event (AE) | Day 1 to End of Trial (Maximum 57 Days from First Dose)
  An AE is defined as any untoward medical occurrence in a clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Part A - Single Dose: Number of Participants with Markedly Abnormal Vital Sign Measurements | Baseline to End of Trial (Maximum 126 Days from First Dose)
  Vital signs will be obtained prior to PK blood draws. Vital signs will include systolic and diastolic blood pressure, heart rate, and body temperature.
Part A - Multiple Dose: Number of Participants with Markedly Abnormal Vital Sign Measurements | Baseline to End of Trial (Maximum 169 Days from First Dose)
  Vital signs will be obtained prior to PK blood draws. Vital signs will include systolic and diastolic blood pressure, heart rate, and body temperature.
Part B: Number of Participants with Markedly Abnormal Vital Sign Measurements | Baseline to End of Trial (Maximum 57 Days from First Dose)
  Vital signs will be obtained prior to PK blood draws. Vital signs will include systolic and diastolic blood pressure, heart rate, and body temperature.
Part A - Single Dose: Number of Participants with Markedly Abnormal Electrocardiograms (ECGs) Results | Baseline to End of Trial (Maximum 126 Days from First Dose)
  Standard 12-lead ECGs will be collected in triplicate (5 minutes apart). The ECGs will be collected prior to PK blood draws and after vital signs at the nominal time points, where applicable.
Part A - Multiple Dose: Number of Participants with Markedly Abnormal Electrocardiograms (ECGs) Results | Baseline to End of Trial (Maximum 169 Days from First Dose)
  Standard 12-lead ECGs will be collected in triplicate (5 minutes apart). The ECGs will be collected prior to PK blood draws and after vital signs at the nominal time points, where applicable.
Part B: Number of Participants with Markedly Abnormal Electrocardiograms (ECGs) Results | Baseline to End of Trial (Maximum 57 Days from First Dose)
  Standard 12-lead ECGs will be collected in triplicate (5 minutes apart). The ECGs will be collected prior to PK blood draws and after vital signs at the nominal time points, where applicable.
Part A - Single Dose: Number of Participants with Markedly Abnormal Clinical Laboratory Results | Baseline to End of Trial (Maximum 126 Days from First Dose)
  Clinical Laboratory Monitoring includes serum chemistry, hematology and urinalysis.
Part A - Multiple Dose: Number of Participants with Markedly Abnormal Clinical Laboratory Results | Baseline to End of Trial (Maximum 169 Days from First Dose)
  Clinical Laboratory Monitoring includes serum chemistry, hematology and urinalysis.
Part B: Number of Participants with Markedly Abnormal Clinical Laboratory Results | Baseline to End of Trial (Maximum 57 Days from First Dose)
  Clinical Laboratory Monitoring includes serum chemistry, hematology and urinalysis.
Part A - Single Dose: Change from Baseline in Serum Prolactin | Baseline to End of Trial (Maximum 126 Days from First Dose)
Part A - Multiple Dose: Change from Baseline in Serum Prolactin | Baseline to End of Trial (Maximum 169 Days from First Dose)
Part B: Change from Baseline in Serum Prolactin | Baseline to End of Trial (Maximum 57 Days from First Dose)
Part A - Single Dose: Number of Participants with Markedly Abnormal Physical Examination Results | Baseline to End of Trial (Maximum 126 Days from First Dose)
Part A - Multiple Dose: Number of Participants with Markedly Abnormal Physical Examination Results | Baseline to End of Trial (Maximum 169 Days from First Dose)
Part B: Number of Participants with Markedly Abnormal Physical Examination Results | Baseline to End of Trial (Maximum 57 Days from First Dose)
Part A - Single Dose: Visual Analog Scale (VAS) Scores for Injection Site Pain Perception | Day 1 immediately post-dose, 1 hour post-dose (+/- 15 minutes), Day 14 and Day 29
  VAS scores at Day 1 immediately post-dose, 1 hour post-dose (+/- 15 minutes), Day 14 and Day 29. The VAS is a test to assess injection site pain. Participants will be asked to give a score between 0-10 to rate pain, with 0 being no pain and 10 being worst possible pain.
Part A - Multiple Dose: Visual Analog Scale (VAS) Scores for Injection Site Pain Perception | 1-hour post-dose Day 1, Day 29, Day 57, Day 85, Day 113
  VAS scores at 1-hour post-dose on Day 1, Day 29, Day 57, Day 85, Day 113. The VAS is a test to assess injection site pain. Participants will be asked to give a score between 0-10 to rate pain, with 0 being no pain and 10 being worst possible pain.
Part B: Visual Analog Scale (VAS) Scores for Injection Site Pain Perception | Day 1 immediately post-dose, 1 hour post-dose (+/- 15 minutes), Day 14 and Day 29
  VAS scores at Day 1 immediately post-dose, 1 hour post-dose (+/- 15 minutes), Day 14 and Day 29. The VAS is a test to assess injection site pain. Participants will be asked to give a score between 0-10 to rate pain, with 0 being no pain and 10 being worst possible pain.
Part A - Single Dose: Change from Baseline of Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline to End of Trial (Maximum 126 Days from First Dose)
  Suicidality will be monitored throughout the trial using the C-SSRS (Columbia-Suicide Severity Rating Scale). This scale consists of a baseline evaluation that assesses the lifetime experience of the subject with suicide events and suicidal ideation and a post-baseline evaluation that focuses on suicidality since the last assessment.The Baseline/Screening Version and the Since Last Visit version of the C-SSRS will be completed by trained trial site staff at each visit. A numerical score will correspond to one of ten categories relating to suicidal ideation and suicidal behavior. A higher score indicates a higher risk of suicidal behavior, but an answer of 'yes' to any question indicates some risk.
Part A - Multiple Dose: Change from Baseline of Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline to End of Trial (Maximum 169 Days from First Dose)
  Suicidality will be monitored throughout the trial using the C-SSRS (Columbia-Suicide Severity Rating Scale). This scale consists of a baseline evaluation that assesses the lifetime experience of the subject with suicide events and suicidal ideation and a post-baseline evaluation that focuses on suicidality since the last assessment.The Baseline/Screening Version and the Since Last Visit version of the C-SSRS will be completed by trained trial site staff at each visit. A numerical score will correspond to one of ten categories relating to suicidal ideation and suicidal behavior. A higher score indicates a higher risk of suicidal behavior, but an answer of 'yes' to any question indicates some risk.
Part B: Change from Baseline of Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline to End of Trial (Maximum 57 Days from First Dose)
  Suicidality will be monitored throughout the trial using the C-SSRS (Columbia-Suicide Severity Rating Scale). This scale consists of a baseline evaluation that assesses the lifetime experience of the subject with suicide events and suicidal ideation and a post-baseline evaluation that focuses on suicidality since the last assessment.The Baseline/ Screening Version and the Since Last Visit version of the C-SSRS will be completed by trained trial site staff at each visit. A numerical score will correspond to one of ten categories relating to suicidal ideation and suicidal behavior. A higher score indicates a higher risk of suicidal behavior, but an answer of 'yes' to any question indicates some risk.
Part A - Single Dose: Number of Injection Site Related Adverse Events | End of Trial (Maximum 126 Days from First Dose)
  An AE is defined as any untoward medical occurrence in a clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.The injection site will be monitored by the investigator to assess the safety and tolerability of the drug.
Part A - Multiple Dose: Number of Injection Site Related Adverse Events | End of Trial (Maximum 169 Days from First Dose)
  An AE is defined as any untoward medical occurrence in a clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.The injection site will be monitored by the investigator to assess the safety and tolerability of the drug.
Part B: Number of Injection Site Related Adverse Events | End of Trial (Maximum 57 Days from First Dose)
  An AE is defined as any untoward medical occurrence in a clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.The injection site will be monitored by the investigator to assess the safety and tolerability of the drug.
Part A - Single Dose: Change from Baseline in Assessment of Extrapyramidal Symptoms (EPS) | Day 1 (predose) to End of Trial (Maximum 126 Days from First Dose)
  EPS will be assessed using Simpson-Angus Scale (SAS), Abnormal Involuntary Movement Scale (AIMS) and Barnes Akathisia Rating Scale (BARS). The SAS consists of a list of 10 symptoms of Parkinsonism. Each item will be rated on a 5-point scale, with a score of 1 representing absence of symptoms and a score of 5 representing a severe condition. The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Each item will be rated on a 5-point scale, with a score of 0 representing absence of symptoms, and a score of 4 indicating a severe condition. The BARS consist of 4 items related to akathisia. The first 3 items will be rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation will be made on a 6-point scale, with 0 representing absence of symptoms and 5 representing severe akathisia.
Part A - Multiple Dose: Change from Baseline in Assessment of Extrapyramidal Symptoms (EPS) | Day 1 (predose) to End of Trial (Maximum 169 Days from First Dose)
  EPS will be assessed using Simpson-Angus Scale (SAS), Abnormal Involuntary Movement Scale (AIMS) and Barnes Akathisia Rating Scale (BARS). The SAS consists of a list of 10 symptoms of Parkinsonism. Each item will be rated on a 5-point scale, with a score of 1 representing absence of symptoms and a score of 5 representing a severe condition. The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Each item will be rated on a 5-point scale, with a score of 0 representing absence of symptoms, and a score of 4 indicating a severe condition. The BARS consist of 4 items related to akathisia. The first 3 items will be rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation will be made on a 6-point scale, with 0 representing absence of symptoms and 5 representing severe akathisia.
Part B: Change from Baseline in Assessment of Extrapyramidal Symptoms (EPS) | Day 1 (predose) to End of Trial (Maximum 57 Days from First Dose)
  EPS will be assessed using Simpson-Angus Scale (SAS), Abnormal Involuntary Movement Scale (AIMS) and Barnes Akathisia Rating Scale (BARS). The SAS consists of a list of 10 symptoms of Parkinsonism. Each item will be rated on a 5-point scale, with a score of 1 representing absence of symptoms and a score of 5 representing a severe condition.
  The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Each item will be rated on a 5-point scale, with a score of 0 representing absence of symptoms, and a score of 4 indicating a severe condition. The BARS consist of 4 items related to akathisia. The first 3 items will be rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation will be made on a 6-point scale, with 0 representing absence of symptoms and 5 representing severe akathisia.
Part A - Single Dose: Change from Baseline in Positive and Negative Syndrome Scale Rating Criteria (PANSS) Score | Baseline to End of Trial (Maximum 126 Days from First Dose)
  The PANSS will be administered using the Structured Clinical Interview-PANSS. The PANSS consists of 3 subscales containing a total of 30 symptom constructs.13 For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. This analysis will include participants with schizophrenia only.
Part A - Multiple Dose: Change from Baseline in Positive and Negative Syndrome Scale Rating Criteria (PANSS) Score | Baseline to End of Trial (Maximum 169 Days from First Dose)
  The PANSS will be administered using the Structured Clinical Interview-PANSS. The PANSS consists of 3 subscales containing a total of 30 symptom constructs.13 For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. This analysis will include participants with schizophrenia only.
Part B: Change from Baseline in Positive and Negative Syndrome Scale Rating Criteria (PANSS) Score | Baseline to End of Trial (Maximum 57 Days from First Dose)
  The PANSS will be administered using the Structured Clinical Interview-PANSS. The PANSS consists of 3 subscales containing a total of 30 symptom constructs.13 For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. This analysis will include participants with schizophrenia only.
Part A - Single Dose: Change from Baseline in Clinical Global Impression-Severity (CGI-S) Score | Baseline to End of Trial (Maximum 126 Days from First Dose)
  The CGI-S Scale will be used to rate the severity of illness for each participant. The scale is a 7-point likert scale, where 1 indicates no illness and 7 indicates extremely ill.
Part A - Multiple Dose: Change from Baseline in Clinical Global Impression-Severity (CGI-S) Score | Baseline to End of Trial (Maximum 169 Days from First Dose)
  The CGI-S Scale will be used to rate the severity of illness for each participant. The scale is a 7-point likert scale, where 1 indicates no illness and 7 indicates extremely ill.
Part B: Change from Baseline in Clinical Global Impression-Severity (CGI-S) Score | Baseline to End of Trial (Maximum 57 Days from First Dose)
  The CGI-S Scale will be used to rate the severity of illness for each participant. The scale is a 7-point likert scale, where 1 indicates no illness and 7 indicates extremely ill.
Part A - Single Dose: Change from Baseline in Subjective Well-being under Neuroleptic Treatment-Short Form (SWN-S) Score | Baseline to End of Trial (Maximum 126 Days from First Dose)
  The subject's feeling of their own well-being will be assessed using the 20 question SWN-S. The questionnaire consists of 20 items and 5 subscales (mental functioning, social integration, emotional regulation, physical functioning, self-control) whose items follow in random order. For items marked with a '+', response choices and scoring are as follows: not at all = 1, hardly at all = 2, a little = 3, somewhat = 4, much = 5, very much = 6. For items marked with a '-', the scoring is reversed; response choices and scoring are as follows: not at all = 6, hardly at all = 5, a little = 4, somewhat = 3, much = 2, very much = 1.
Part A - Multiple Dose: Change from Baseline in Subjective Well-being under Neuroleptic Treatment-Short Form (SWN-S) Score | Baseline to End of Trial (Maximum 169 Days from First Dose)
  The subject's feeling of their own well-being will be assessed using the 20 question SWN-S. The questionnaire consists of 20 items and 5 subscales (mental functioning, social integration, emotional regulation, physical functioning, self-control) whose items follow in random order. For items marked with a '+', response choices and scoring are as follows: not at all = 1, hardly at all = 2, a little = 3, somewhat = 4, much = 5, very much = 6. For items marked with a '-', the scoring is reversed; response choices and scoring are as follows: not at all = 6, hardly at all = 5, a little = 4, somewhat = 3, much = 2, very much = 1.
Part B: Change from Baseline in Subjective Well-being under Neuroleptic Treatment-Short Form (SWNS) Score | Baseline to End of Trial (Maximum 57 Days from First Dose)
  The subject's feeling of their own well-being will be assessed using the 20 question SWN-S. The questionnaire consists of 20 items and 5 subscales (mental functioning, social integration, emotional regulation, physical functioning, self-control) whose items follow in random order. For items marked with a '+', response choices and scoring are as follows: not at all = 1, hardly at all = 2, a little = 3, somewhat = 4, much = 5, very much = 6. For items marked with a '-', the scoring is reversed; response choices and scoring are as follows: not at all = 6, hardly at all = 5, a little = 4, somewhat = 3, much = 2, very much = 1.
Part A - Single Dose: Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score | Baseline to End of Trial (Maximum 126 Days from First Dose)
  The MADRS will be utilized as the primary assessment of a subject's level of depressive symptoms and must be administered using a structured interview guide. This scale consists of 10 items each with 7 defined grades of severity.This analysis will include participants with bipolar only.
Part A - Multiple Dose: Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score | Baseline to End of Trial (Maximum 169 Days from First Dose)
  The MADRS will be utilized as the primary assessment of a subject's level of depressive symptoms and must be administered using a structured interview guide. This scale consists of 10 items each with 7 defined grades of severity.This analysis will include participants with bipolar only.
Part B: Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score | Baseline to End of Trial (Maximum 57 Days from First Dose)
  The MADRS will be utilized as the primary assessment of a subject's level of depressive symptoms and must be administered using a structured interview guide. This scale consists of 10 items each with 7 defined grades of severity. This analysis will include participants with bipolar only.
Part A - Single Dose: Change from Baseline in Young Mania Rating Scale (YMRS) Score | Baseline to End of Trial (Maximum 126 Days from First Dose)
  The YMRS consists of 11 items assessing the core symptoms of mania and is based on the subject's subjective report of his or her clinical condition. Each item has 5 defined categories of severity with 4 items graded on a 0 to 8 scale (irritability, speech, content, and disruptive-aggressive behavior) and 7 items graded on a 0 to 4 scale. This analysis will include participants with bipolar only.
Part A - Multiple Dose: Change from Baseline in Young Mania Rating Scale (YMRS) Score | Baseline to End of Trial (Maximum 169 Days from First Dose)
  The YMRS consists of 11 items assessing the core symptoms of mania and is based on the subject's subjective report of his or her clinical condition. Each item has 5 defined categories of severity with 4 items graded on a 0 to 8 scale (irritability, speech, content, and disruptive-aggressive behavior) and 7 items graded on a 0 to 4 scale. This analysis will include participants with bipolar only.
Part B: Change from Baseline in Young Mania Rating Scale (YMRS) Score | Baseline to End of Trial (Maximum 57 Days from First Dose)
  The YMRS consists of 11 items assessing the core symptoms of mania and is based on the subject's subjective report of his or her clinical condition. Each item has 5 defined categories of severity with 4 items graded on a 0 to 8 scale (irritability, speech, content, and disruptive-aggressive behavior) and 7 items graded on a 0 to 4 scale. This analysis will include participants with bipolar only.
Part A - Single Dose: Change from Baseline in Clinical Global Impression-Bipolar Version (CGI-BP) Score | Baseline to End of Trial (Maximum 126 Days from First Dose)
  Severity of illness will be measured using the CGI-BP score. To assess CGI-S, the investigator will answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the subject at this time?" Response choices include: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill subjects. This analysis will include participants with bipolar only.
Part A - Multiple Dose: Change from Baseline in Clinical Global Impression-Bipolar Version (CGI-BP) Score | Baseline to End of Trial (Maximum 169 Days from First Dose)
  Severity of illness will be measured using the CGI-BP score. To assess CGI-S, the investigator will answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the subject at this time?" Response choices include: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill subjects. This analysis will include participants with bipolar only.
Part B: Change from Baseline in Clinical Global Impression-Bipolar Version (CGI-BP) Score | Baseline to End of Trial (Maximum 57 Days from First Dose)
  Severity of illness will be measured using the CGI-BP score. To assess CGI-S, the investigator will answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the subject at this time?" Response choices include: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill subjects. This analysis will include participants with bipolar only.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Woodland International Research Group, Little Rock, Arkansas
  - Collaborative Neuroscience Network, Garden Grove, California
  - Hassman Research Institute, Berlin, New Jersey
  - Community Clinical Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com